CLINICAL TRIAL: NCT06742723
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Event-driven Study to Assess the Efficacy, Safety and Tolerability of Baxdrostat in Combination With Dapagliflozin Compared With Dapagliflozin Alone on Renal Outcomes and Cardiovascular Mortality in Participants With Chronic Kidney Disease and High Blood Pressure
Brief Title: A Phase III Renal Outcomes and Cardiovascular Mortality Study to Investigate the Efficacy and Safety of Baxdrostat in Combination With Dapagliflozin in Participants With Chronic Kidney Disease and High Blood Pressure
Acronym: BaxDuo-Pacific
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6972C00002; 2023-506460-14-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease and Hypertension
Keywords: Chronic kidney disease; Hypertension; Blood pressure; Baxdrostat; Dapagliflozin; Event-Driven; Outcome
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: International, multi-centre, randomised, double-blind, parallel-group, placebo-controlled, event-driven, outcome
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baxdrostat/dapagliflozin (Experimental): Participants randomised to the baxdrostat/dapagliflozin arm will initially receive a lower dose of baxdrostat and standard dose dapagliflozin. For participants that meet the up-titration criteria, baxdrostat may be up-titrated to higher dose.
  Interventions: Drug: Baxdrostat/dapagliflozin
- Placebo/dapagliflozin (Placebo Comparator): Patients will receive one dose of dapagliflozin comparator in combination with matching placebo daily.
  Interventions: Drug: Placebo/dapagliflozin

INTERVENTIONS:
Drug: Baxdrostat/dapagliflozin — baxdrostat tablet
  dapagliflozin tablet
  Other Names: Baxdrostat CIN-107
  Arms: Baxdrostat/dapagliflozin
Drug: Placebo/dapagliflozin — dapagliflozin tablet
  placebo tablet
  Arms: Placebo/dapagliflozin

SUMMARY:
International, Multicenter, Double-Blind, Placebo-Controlled and Event-driven study to assess efficacy, safety and Tolerability of Baxdrostat in combination with Dapagliflozin on renal outcomes and cardiovascular mortality in participants with chronic kidney disease and high blood pressure

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy, safety, and tolerability of baxdrostat in combination with dapagliflozin, compared with placebo and dapagliflozin, in reducing the risk of the composite endpoint of ≥ 50% sustained decline in eGFR, kidney failure, HF events, or CV death in participants with CKD and HTN.

This study consists of a 4-week dapagliflozin Run-in Period for participants untreated with SGLT2i at screening, and a double-blinded period where participants will receive either baxdrostat/dapagliflozin or placebo/dapagliflozin.

Site visits will take place at 2-, 4-, 8-, 16-, 34, and 52-weeks following randomisation. Thereafter visits will occur approximately every 4 months.

The study closure procedures will be initiated when the predetermined number of primary endpoint events is predicted to have occurred (N = 845) ie, the PACD. All randomised participants including any participants who have prematurely discontinued study intervention will be scheduled for a SCV within 6 weeks of the PACD. This period can be extended by AstraZeneca.

In case of premature discontinuation of blinded study intervention, participants will continue in the study and receive dapagliflozin 10 mg, unless the participant meets dapagliflozin specific discontinuation criteria. Baxdrostat/placebo should not be administered without dapagliflozin: baxdrostat/placebo should be interrupted if dapagliflozin is interrupted (baxdrostat/placebo may be resumed with dapagliflozin, if dapagliflozin is resumed), and should be permanently discontinued if dapagliflozin is permanently discontinued. If study intervention is temporarily or permanently discontinued, the participant should remain in the study, and it is important that the scheduled study visits (including the PTDV for participants with permanent discontinuation of study intervention) and data collection continue according to the study protocol until the SCV.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of any sex and gender must be ≥ 18 years of age at the time of signing the informed consent.
2. Participants with (a) or (b):

   a) eGFR 30-59 mL/min/1.73 m² (local or central laboratory value) AND:
   * UACR ≥ 30 mg/g (3.39 mg/mmol) and < 500 mg/g (56.5 mg/mmol) (central laboratory value only), or
   * UACR ≥ 500 mg/g (56.5 mg/mmol) and ≤ 5000 mg/g (565 mg/mmol) (local or central laboratory value), or
   * UPCR ≥ 700 mg/g (79 mg/mmol) and ≤ 7000 mg/g (790 mg/mmol) (local laboratory value only).

     (b) eGFR 60-75 mL/min/1.73 m² (local or central laboratory value) AND:
   * UACR ≥ 500 mg/g (56.5 mg/mmol) ) and ≤ 5000 mg/g (565 mg/mmol) (local or central laboratory value), or
   * UPCR ≥ 700 mg/g (79 mg/mmol) and ≤ 7000 mg/g (790 mg/mmol) (local laboratory value only)
3. [obsolete]
4. Participants with history of HTN and a SBP ≥ 130 mmHg (the most recent value within 4 weeks prior to screening or at the Screening Visit) and ≥ 120 mmHg at the Randomisation Visit.
5. Stable and maximum tolerated dose of an ACEi or an ARB (not both) for at least 4 weeks prior to Screening Visit.
6. Participants with:

   1. Serum or plasma potassium ≥ 3.0 and ≤ 4.8 mmol/L if eGFR ≥ 45 mL/min/1.73 m2 (local or central laboratory values)
   2. Serum or plasma potassium ≥ 3.0 and ≤ 4.5 mmol/L if eGFR < 45 mL/min/1.73 m2 (local or central laboratory values)

Exclusion Criteria:

1. Systolic blood pressure > 180 mmHg, or diastolic BP > 110 mmHg at screening.
2. Known hyperkalaemia, defined as potassium of ≥ 5.5 mmol/L within 3 months at screening.
3. Serum sodium < 135 mmol/L (central or local laboratory values obtained within 4 weeks prior to screening or at the Screening Visit).

4. Participants with T1DM will be excluded, except:

1. For US only: patients with T1DM treated with SGLT2i for at least 4 months, without DKA during that period, and who have experience with ketone monitoring are eligible for inclusion.
2. For Japan only: patients with T1DM treated with dapagliflozin 10 mg for at least 4 months, without DKA during the period of dapagliflozin treatment are eligible for inclusion.

   5 Uncontrolled T2DM with HbA1c > 10.5% (> 91 mmol/mol) (central or local laboratory values obtained within 3 months prior to screening or at the Screening Visit).

   6 New York Heart Association functional HF class IV at screening.

   7 Stroke, transient ischaemic cerebral attack, valve implantation or valve replacement, carotid surgery, or carotid angioplasty, acute coronary syndrome, or hospitalisation for worsening heart failure within previous 3 months prior to randomisation.

   8 Documented history of adrenal insufficiency.

   9 Any dialysis (including for acute kidney injury) within 3 months prior to Screening Visit.

   10 Any acute kidney injury within 3 months prior to the Screening Visit.

   11 History of organ transplant or bone marrow transplant, or planned organ transplant within 6 months following randomisation (including kidney transplant).

   12 Any clinical condition requiring systemic immunosuppression therapy other than maintenance therapy (stable for at least 3 months prior to Visit 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2029-12-18 (Estimated); Study Completion 2029-12-18 (Estimated)

PRIMARY OUTCOMES:
To determine if baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of the composite endpoint of ≥ 50% sustained decline in eGFR, kidney failure, Heart Failure events(HF), or CV death. | Up to 37 months
  Time to the first occurrence of any of the components of the composite of:
  Kidney disease progression
  * ≥ 50% sustained decline in eGFR
  * Onset of kidney failure:
    * Sustained eGFR < 15 mL/min/1.73 m2 or
    * Chronic dialysis treatment or
    * Receiving a kidney transplant or
    * Death with a renal primary cause (death due to kidney failure when dialysis is not given)
  CV events
  * HF with or without hospitalisation
  * CV death

SECONDARY OUTCOMES:
To determine if baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of the composite endpoint of ≥ 50% sustained decline in eGFR, kidney failure or CV death. | Up to 37 months
  To determine if baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of the composite endpoint of ≥ 50% sustained decline in eGFR, kidney failure, or CV death.
To determine whether baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of the composite endpoint of kidney failure | Up to 37 months
  Time to the first occurrence of any of the components of the composite of:
  • Onset of kidney failure:
  * Sustained eGFR < 15 mL/min/1.73 m2 or
  * Chronic dialysis treatment or
  * Receiving a kidney transplant or
  * Death with a renal primary cause (death due to kidney failure when dialysis is not given)
To determine whether baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of MACE (Major Adverse Cardiac Events). | Up to 37 months
  Time to the first occurrence of any of the components of the composite of: CV (cardiovascular) death, HF (heart failure) with and without hospitalization, Myocardial Infraction, Stroke
To determine whether baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of the composite endpoint of CV (cardiovascular) death. | Up to 37 months
  Time to the first occurrence of any of the components of the composite of CV (cardiovascular) death
To determine whether baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of the composite endpoint of all-cause death. | Up to 37 months
  Time to the first occurrence of any of the components of the composite of all-cause death

OTHER OUTCOMES:
To assess the safety and tolerability of baxdrostat/dapagliflozin compared with placebo/dapagliflozin. | Up to 37 months
  Safety and tolerability will be evaluated in terms of the following endpoints:
  * Occurrence and time to first occurrence of AEs, SAEs, SAEs with outcome death, DAEs, possibly related AEs as assessed by Investigator.
  * Observed values, change from baseline and time to first treatment-emergent abnormality in laboratory parameters.
  * Observed values, change from baseline and time to first treatment-emergent abnormality in vital signs, ECG.
  * Occurrence and time to first occurrence of AESIs: hyperkalaemia, hyponatraemia, and hypotension events that require medical intervention. -Exposure to study treatment will be described

CONTACTS AND LOCATIONS:
Locations (586):
- United States (114):
  - Research Site, Fairhope, Alabama
  - Research Site, Surprise, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Canoga Park, California
  - Research Site, Concord, California
  - Research Site, Fremont, California
  - Research Site, Fullerton, California
  - Research Site, Inglewood, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, Tarzana, California
  - Research Site, Arvada, Colorado
  - Research Site, Denver, Colorado
  - Research Site, New Britain, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Lake City, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Riverview, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Austell, Georgia
  - Research Site, Brunswick, Georgia
  - Research Site, Conyers, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Riverdale, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Champaign, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Hutchinson, Kansas
  - Research Site, Kansas City, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Kenner, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, West Monroe, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, New Bedford, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Garden City, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Norfolk, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Eatontown, New Jersey
  - Research Site, Albany, New York
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Sanford, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Bridgeville, Pennsylvania
  - Research Site, Butler, Pennsylvania
  - Research Site, Exton, Pennsylvania
  - Research Site, Media, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Humble, Texas
  - Research Site, Lewisville, Texas
  - Research Site, Pasadena, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Arlington, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Woodbridge, Virginia
  - Research Site, Seattle, Washington
- Argentina (13):
  - Research Site, CABA
  - Research Site, Ciudad Autonoma de Bs As
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Lanús
  - Research Site, Lanús Este
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, San Nicolás
  - Research Site, Santa Fe
  - Research Site, Santiago del Estero
  - Research Site, Temperley
- Australia (8):
  - Research Site, Adelaide
  - Research Site, Darlinghurst
  - Research Site, Elizabeth Vale
  - Research Site, Gosford
  - Research Site, Perth
  - Research Site, Southport
  - Research Site, St Leonards
  - Research Site, Wollongong
- Belgium (14):
  - Research Site, Aalst
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Hasselt
  - Research Site, Ieper
  - Research Site, Jette
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mechelen
  - Research Site, Namur
  - Research Site, Roeselare
  - Research Site, Ronse
  - Research Site, Sint-Truiden
- Brazil (13):
  - Research Site, Barretos
  - Research Site, Belém
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Joinville
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (16):
  - Research Site, Byala
  - Research Site, Dupnitsa
  - Research Site, Gabrovo
  - Research Site, Gotse Delchev
  - Research Site, Kozloduy
  - Research Site, Lom
  - Research Site, Pernik
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sandanski
  - Research Site, Sevlievo
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Yambol
- Canada (14):
  - Research Site, Edmonton, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Saint John, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Chile (5):
  - Research Site, Araucania
  - Research Site, Santiago
  - Research Site, Valdivia
  - Research Site, Victoria
  - Research Site, Viña del Mar
- China (41):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongwan
  - Research Site, Fuyang
  - Research Site, Guangzhou
  - Research Site, Hefei
  - Research Site, Hengyang
  - Research Site, Huaian
  - Research Site, Jiaxing
  - Research Site, Jilin
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Lanzhou
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Panjin
  - Research Site, Pingxiang
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Wanzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xianyang
  - Research Site, Yantai
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
  - Research Site, Zhongshan
  - Research Site, Zhuzhou
  - Research Site, Zigong
- Colombia (6):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Medellín
  - Research Site, Montería
  - Research Site, Pasto
- Czechia (10):
  - Research Site, Brandýs nad Labem
  - Research Site, Frýdek-Místek
  - Research Site, Jilemnice
  - Research Site, Krnov
  - Research Site, Mladá Boleslav
  - Research Site, Náchod
  - Research Site, Olomouc
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Slaný
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Copenhagen E
  - Research Site, Herlev
  - Research Site, Herning
  - Research Site, Holbæk
  - Research Site, Kolding
- Egypt (3):
  - Research Site, Alexandria
  - Research Site, Cairo
  - Research Site, Dakahlia
- France (24):
  - Research Site, Amiens
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, La Roche-sur-Yon
  - Research Site, Le Mans
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Quimper
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
- Germany (28):
  - Research Site, Bad Homburg
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Brandenburg
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Friedrichsthal
  - Research Site, Görlitz
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Herne
  - Research Site, Karlsburg
  - Research Site, Karlsruhe
  - Research Site, Landshut
  - Research Site, Mainz
  - Research Site, Obertshausen
  - Research Site, Offenbach
  - Research Site, Potsdam
  - Research Site, Reinfeld (Holstein)
  - Research Site, Rostock
  - Research Site, Rotenburg (Wümme)
  - Research Site, Stuttgart
  - Research Site, Ulm
  - Research Site, Wermsdorf
  - Research Site, Zwenkau
- Greece (6):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (10):
  - Research Site, Budapest
  - Research Site, Dunaújváros
  - Research Site, Encs
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Nyíregyháza
  - Research Site, Szeged
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg
- India (9):
  - Research Site, Bangalore
  - Research Site, Belagavi
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Vijayawada
- Israel (11):
  - Research Site, Afula
  - Research Site, Ashdod
  - Research Site, Be’er Ya‘aqov
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Tiberias
- Italy (16):
  - Research Site, Bassano del Grappa
  - Research Site, Bologna
  - Research Site, Desio
  - Research Site, Foggia
  - Research Site, Genoa
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Pordenone
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Torino
  - Research Site, Tradate
- Japan (52):
  - Research Site, Aira
  - Research Site, Amagasaki-shi
  - Research Site, Beppu-shi
  - Research Site, Chigasaki-shi
  - Research Site, Fujinomiya-shi
  - Research Site, Hakodate-shi
  - Research Site, Hamamatsu
  - Research Site, Higashihiroshima-shi
  - Research Site, Iizuka-shi
  - Research Site, Inashiki-gun
  - Research Site, Itabashi-ku
  - Research Site, Iwata-shi
  - Research Site, Kagoshima
  - Research Site, Kamakura-shi
  - Research Site, Kanazawa
  - Research Site, Kashiwara-shi
  - Research Site, Kasugai-shi
  - Research Site, Kita-ku
  - Research Site, Kitakyushu
  - Research Site, Kitakyushu-shi
  - Research Site, Kobe
  - Research Site, Kumagaya-shi
  - Research Site, Kurashiki Shi
  - Research Site, Kuse-gun
  - Research Site, Kuwana-shi
  - Research Site, Kyoto
  - Research Site, Matsusaka-shi
  - Research Site, Matsuyama
  - Research Site, Meguro-ku
  - Research Site, Minatoku
  - Research Site, Minokamo Shi
  - Research Site, Miyakonojo-shi
  - Research Site, Morioka
  - Research Site, Nagaoka-shi
  - Research Site, Naka
  - Research Site, Narita-shi
  - Research Site, Obihiro-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Ōme
  - Research Site, Ōmihachiman
  - Research Site, Saga
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shibuya-ku
  - Research Site, Tanabe-shi
  - Research Site, Toyoake-shi
  - Research Site, Toyohashi
  - Research Site, Tsu
  - Research Site, Yaizu-shi
  - Research Site, Yokohama
  - Research Site, Yoshida-gun
- Malaysia (8):
  - Research Site, Ampang
  - Research Site, Cheras
  - Research Site, Ipoh
  - Research Site, Kajang
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Site, Seremban
  - Research Site, Seri Manjung
- Mexico (10):
  - Research Site, Chihuahua City
  - Research Site, Cuauhtémoc
  - Research Site, D.F
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Mazatlán
  - Research Site, Mérida
  - Research Site, San Luis Potosí City
  - Research Site, Veracruz
  - Research Site, Zapopan
- Netherlands (9):
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Dordrecht
  - Research Site, Groningen
  - Research Site, Hilversum
  - Research Site, Leiden
  - Research Site, Maastricht
  - Research Site, Nieuwegein
  - Research Site, Zwolle
- Peru (5):
  - Research Site, Arequipa
  - Research Site, Bellavista
  - Research Site, Chorrillos
  - Research Site, Lima
  - Research Site, Piura
- Philippines (8):
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Laguna
  - Research Site, Manadaluyong City
  - Research Site, Manila
  - Research Site, Quezon City
  - Research Site, San Fernando City
- Poland (18):
  - Research Site, Bialystok
  - Research Site, Gdynia
  - Research Site, Gmina Świecie
  - Research Site, Jasło
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Piaseczno
  - Research Site, Poznan
  - Research Site, Pruszków
  - Research Site, Radom
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Tczew
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Żywiec
- Romania (7):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Oradea
  - Research Site, Suceava
  - Research Site, Timișoara
- Saudi Arabia (4):
  - Research Site, Al-Ahsa
  - Research Site, Dammam
  - Research Site, Riyadh
  - Research Site, Riyadh/MENA
- Serbia (5):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Sad
- Research Site, Singapore, Singapore
- Slovakia (9):
  - Research Site, Košice
  - Research Site, Kráľovský Chlmec
  - Research Site, Myjava
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Púchov
  - Research Site, Trenčín
  - Research Site, Trnava
  - Research Site, Žilina
- South Africa (11):
  - Research Site, Bellville
  - Research Site, Benoni
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Extension 8, Lenasia
  - Research Site, KwaDukuza
  - Research Site, Lenasia
  - Research Site, Midrand
  - Research Site, Newton
  - Research Site, Parow
- South Korea (10):
  - Research Site, Ansan-si
  - Research Site, Anyang-si
  - Research Site, Busan
  - Research Site, Cheonan-si
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Wŏnju
  - Research Site, Yangsan
- Spain (10):
  - Research Site, A Coruña
  - Research Site, Almería
  - Research Site, Badalona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Palma deMallorca
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (6):
  - Research Site, Danderyd
  - Research Site, Huddinge
  - Research Site, Karlstad
  - Research Site, Linköping
  - Research Site, Uppsala
  - Research Site, Vaxjo
- Taiwan (5):
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yung Kang City
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Banphaeo
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Mueang
  - Research Site, Phutthamonthon
  - Research Site, Ubonratchathani
- Turkey (Türkiye) (10):
  - Research Site, Adana
  - Research Site, Adapazarı
  - Research Site, Altındağ
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Haliliye
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
  - Research Site, Şahinbey
- Ukraine (7):
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zhytomyr
- United Kingdom (11):
  - Research Site, Bradford
  - Research Site, Bristol
  - Research Site, Canterbury
  - Research Site, Cardiff
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Hownslow
  - Research Site, London
  - Research Site, Salford
  - Research Site, Southampton
  - Research Site, Swansea
- Vietnam (5):
  - Research Site, Da Nang
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Rach Gia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Dwyer JP, Maklad N, Vedin O, Monyak J, Myte R, Chertow GM, Heerspink HJL, Little DJ. Efficacy and Safety of Baxdrostat in Participants with CKD and Uncontrolled Hypertension: A Randomized, Double-Blind, Placebo-Controlled Trial. J Am Soc Nephrol. 2025 Sep 6. doi: 10.1681/ASN.0000000849. Online ahead of print. No abstract available. PMID 40913594